CLINICAL TRIAL: NCT03960151
Title: Phase II Study of Rolapitant Plus Olanzapine, Palonosetron, and Dexamethasone in Patients With Germ Cell Tumors Undergoing 5-day Cisplatin-based Chemotherapy.
Brief Title: Rolapitant Plus Olanzapine in Multiday Cisplatin Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Compound was sold by funder and development ceased.
Sponsor: Costantine Albany (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Costantine Albany, Sponsor Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU16-254
Record Dates: First submitted 2018-03-26; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — rolapitant; Palonosetron; Olanzapine; Dexamethasone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rolapitant (Experimental): Rolapitant plus Olanzapine, Palonosetron, and Dexamethasone
  Interventions: Drug: Rolapitant; Drug: Palonosetron; Drug: Olanzapine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Rolapitant — Rolapitant 180mg PO, Days 1 and 5
  Other Names: Varubi
Drug: Palonosetron — Palonosetron 0.25 mg IV, Days 1,3, and 5.
  Other Names: Aloxi
Drug: Olanzapine — Olanzapine 10 mg PO PM, Days 2,3,4,5,6-8
  Other Names: Zyprexa
Drug: Dexamethasone — Dexamethasone 20 mg AM, Days 1,2 and 3
  Other Names: steroid

SUMMARY:
Phase II study of Rolapitant plus Olanzapine, Palonosetron, and Dexamethasone in patients with germ cell tumors undergoing 5-day Cisplatin-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 15 years at the time of consent.
* Must be able to take oral medications (swallow pills)
* ECOG Performance Status of 0-2 within 14 days prior to registration.
* Histological or serological confirmation of germ cell tumor planning on receiving a standard 5 day cisplatin based chemotherapy regimen.
* Patients must have had no nausea or vomiting for 24 hours and no antiemetic use for 72 hours prior to starting protocol therapy.
* No active central nervous system (CNS) metastases. Patients with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis. A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic.
* Prior cancer treatments are not allowed. Patients have to be chemotherapy naïve.
* Absolute Neutrophil Count (ANC) ≥ 1 K/mm3
* Hemoglobin (Hgb) ≥ 10 g/dL
* Platelets (Plt) ≥ 100 K/mm3
* Creatinine ≤ 2 mg/dL
* Bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN
* No concurrent use of thioridazine or pimozide. No use of agents expected to induce the metabolism of rolapitant which include: Rifampin, Rifabutin, Phenytoin, Carbamazepine, and Barbiturates.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* Patients and their partners must agree to use a highly effective method of birth control from the signing of the informed consent form until 90 days following the last dose of rolapitant.

Exclusion Criteria:

* Any untreated central nervous system (CNS) metastases.
* Treatment with any investigational drug within 30 days prior to registration.
* Concurrent participation in a clinical trial which involves another investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 8 Days
  Determine the complete response (CR) rate defined as no emesis and no use of rescue medications in germ cell tumor patients treated with rolapitant plus Olanzapine in combination with palonosetron a 5HT3RA and dexamethasone on Cycle 1 Day 1 through Day 8

SECONDARY OUTCOMES:
Complete Response Rate: Acute Phase | 5 Days
  Determine the CR rate in the acute phase (Days 1-5) defined as no emesis and no use of rescue medications in germ cell tumor patients treated with rolapitant plus Olanzapine in combination with palonosetron a 5HT3RA and dexamethasone on Cycle 1 Day 1 through Day 5
Complete Response Rate: Delayed Phase | 2 Days
  Determine the CR rate in the delayed phase (Days 6-8) defined as no emesis and no use of rescue medications in germ cell tumor patients treated with rolapitant plus Olanzapine in combination with palonosetron a 5HT3RA and dexamethasone on Cycle 1 Day 6 through Day 8
Frequency, intensity, and duration of nausea | 8 Days
  Determine the frequency, intensity and duration of nausea on Days 1-8 in Cycle 1. The frequency, intensity and duration of nausea will be captured via daily self-assessment patient logs.
Frequency of vomiting or retching. | 8 Days
  Determine the frequency, intensity and duration of vomiting or retching on Days 1-8 in Cycle 1. The frequency of vomiting and retching will be captured via daily self-assessment patient logs.
Intensity of Vomiting or retching. | 8 Days
  Determine the intensity of vomiting or retching on Days 1-8 in Cycle 1. The intensity of vomiting and retching will be captured via daily self-assessment patient logs.
Duration of Vomiting or retching | 8 Days
  Determine the duration of vomiting or retching on Days 1-8 in Cycle 1. The duration of vomiting and retching will be captured via daily self-assessment patient logs.
Rate of no nausea | 8 Days
  Determine the rate of no nausea defined as < 5mm on a 0-100mm visual analog scale (VAS) on Days 1-5 and Days 6-8 on Cycle 1
Use of rescue medications | 8 Days
  Describe the use of rescue medications as defined in the protocol
Assess adverse events of regimen using CTCAE v4. | 8 Days
  Safety and toxicity will be assessed using CTCAE v4

CONTACTS AND LOCATIONS:
Overall Officials: Costantine Albany, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided